CLINICAL TRIAL: NCT05518955
Title: Strategies Establishment for Promoting Sleep Quality and Quantity of Patients Requiring Intensive Care: Verifying the Effect of Virtual Reality Integrated Into Multicomponent Interventions
Brief Title: VR Integrated Into Multicomponent Interventions for Improving Sleep in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hsiao-Yean Chiu (Other)
Responsible Party: Sponsor-Investigator, Hsiao-Yean Chiu, Associated professor, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202202058
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Critical Care; Sleep Quality
Keywords: Intensive care unit; Sleep deprivation; Virtual reality; multicomponent intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality combine with sleep promotion routine (Experimental): Participants will receive virtual reality for 30 minutes before bedtime then will be placed on an eye mask and combine with the sleep promotion routine. The intervention duration need continues for two days or until discharge from ICU.
  Interventions: Behavioral: Virtual reality and eye mask
- control group (No Intervention): Participants will receive eye masks during their sleep for consecutive two days or until discharge from ICU.

INTERVENTIONS:
Behavioral: Virtual reality and eye mask — Participates will receive a virtual reality program 30 min before their sleep and combine with the sleep routine program for consecutive 2 nights in the ICU.
  Arms: Virtual reality combine with sleep promotion routine

SUMMARY:
Background: The patients who are admitted to ICUs mostly experience sleep disturbance. Seeking an effective strategy and integrating it into the daily routine is of clinical importance. Therefore, we aim to examine the effects of guided virtual reality integrated into the multicomponent program (SLEEP care) on sleep quality and quantity in critically ill patients. This will be a randomized controlled trial with assessor-blinded and two-arm parallel-group design. A total of 120 critical ill adults will be randomly allocated to the SLEEP care group and eyemask groups in a 1:1 ratio (60 participants in each group).

DETAILED DESCRIPTION:
This study is expected to enroll 120 critically ill patients. We will collect basic data on the first day of admission to the intensive care unit, including demographics and disease characteristics, pain, anxiety, and stress, sleep quality and quantity, measure 5-minute HRV, wear an actigraph watch, and connect to the on-lead EEG sensor, and attach the brain wave to monitor the brain wave and sleep cycle. Then they will be randomly assigned 1:1, dividing into SLEEP care group and eyemask group. Participants who are in the control will receive eyemask intervention and daily care in the ICU. Participants who are assigned to the SLEEP care group will receive the VR and night sleep promotion routine. The researcher will assist participants to wear a virtual reality helmet for a 30-minute program at 10 pm, and then remove the helmet and wear eye masks until 6:30 in the morning. The ICU routine care of promoting sleep is still maintained. The next morning (the second day of the ICU), the researcher will assist participants to remove EEG sensors and evaluate the RCSQ scale to understand the previous night's sleep. The above process will repeat for three days (ICU days 1 to 3) until the intervention and measurement during the intensive care unit are completed on the morning of the fourth day. In order to understand the impact of sleep on cognitive function during the stay in the intensive care units and after discharge, the PSQI, VAS of pain, anxiety, and stress (confounders), and MOCA will be evaluated in the first and sixth months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years and above.
* Conscious and able to communicate with Chinese or Mandarin.
* To stay in ICU at least 72 hrs

Exclusion Criteria:

* The medical history of sleep disorder, cognition impairment, psychiatric disorders, seizures, visual difficulty or hearing difficulty
* The APACHE II score over than 25
* The participates who are delirium

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Changes in subjective sleep quality from first day to 3rd day of ICU recruitment | The 1st to 3rd day of ICU recruitment
  Subjective sleep quality in ICU is assessed by Richards-Campbell Sleep Questionnaire(RCSQ). The mean of total score is 0-100. The higher score means the better sleep quality.
Change of subjective sleep quality from before ICU and admission for 30 and 180 days after ICU discharge | The 1st day of ICU recruitment, 30 and 180 days days after ICU discharge
  sleep quality is assessed by Pittsburgh Sleep Quality. Index(PSQI). The total score is 0-21. The higher score means the worse sleep quality.
Change of objective sleep from 1st day to 3rd day of ICU recruitment | The 1st day to 3rd day of ICU recruitment
  Objective sleep quality in ICU is measured by actigraphy

SECONDARY OUTCOMES:
Change of quality of life from the first day of ICU recruitment, 30 and 180 day after ICU discharge | The 30 and 180 days after ICU discharge
  Cognitive function is assessed by MoCA. The total scales is 30. The scale is more than 26 means the patients do not have cognitive impairment.
Delirium occurrence | The 1st to 3th days of ICU recruitment
  Delirium is assessed by Intensive Care Delirium Screening Checklist (ICDSC) or Confusion Assessment Method for the intensive care unit (CAM-ICU)
Change of heart rate variability | The 1st and 3rd days of ICU recruitment
  Heart rate variability is measured by portable ECG recorder and analyzer.
Change from baseline on anxiety | the 1st day of ICU recruitment and up to 30 and 180 days
  Anxiety is assessed by Visual Analog Scale (VAS) anxiety scoring.The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain(score of 10) .The higher score means the very anxiety.
Change of stress | The 1st day of ICU recruitment, 30 and 180 days after ICU discharge
  Stress is assessed by Visual Analog Scale(VAS) stress scoring.The scale is most commonly anchored by "no stress" (score of 0) and "very stressful(score of 10) .The higher score means the very stressful.
Change of pain | The 1st day of ICU recruitment, 30 and 180 days days after ICU discharge
  Pain is assessed by Visual Analog Scale(VAS) pain scoring.The scale is most commonly anchored by "no pain" (score of 0) and "very painful(score of 10) .The higher score means the very painful.
Electroencephalography | The 1st day to 3rd day of ICU recruitment
  Electroencephalography is measured by SOMNOwatch

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yean Chiu, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No